CLINICAL TRIAL: NCT04719897
Title: Effects of Stressful Life Experiences on the Acquisition of a Coping Skill in Adolescents With Elevated Depression Symptoms
Brief Title: Life Experiences in Adolescents and the Development of Skills
Acronym: LEADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rachel Vaughn-Coaxum, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY20040133; 1K23MH123685-01 (NIH)
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Depression in Adolescence; Adverse Childhood Experiences
Keywords: Depression; Adolescents; Cognitive Behavioral Therapy; Childhood Adversity; Cognitive Function; Psychophysiology
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FIRST: Repairing Thoughts (Experimental)
  Interventions: Behavioral: FIRST: Repairing Thoughts

INTERVENTIONS:
Behavioral: FIRST: Repairing Thoughts — This intervention uses the Repairing Thoughts cognitive restructuring module of the FIRST (Feeling Calm, Increasing Motivation, Repairing Thoughts, Solving Problems, Trying the Opposite) cognitive behavioral therapy protocol. This psychotherapy module teaches adolescents that thoughts are linked to feelings and behaviors, and that thoughts are often "guesses" to interpreting the world around us. Adolescents are taught to notice their thoughts in real-time and evaluate the evidence that supports or contradicts the thoughts and interpretation. Adolescents are then taught strategies to re-interpret thoughts in a more realistic manner and notice changes in emotional and behavioral responses. Clinicians are provided with examples to enhance learning, and between-session practice is assigned as "homework."

SUMMARY:
The primary objective of this study is to assess acquisition and retention of a Cognitive Behavioral Therapy (CBT)-based "cognitive restructuring" skill, among young adolescents (12-15 years of age) with elevated depression symptoms and with population-level variability in lifetime exposure to adverse childhood experiences. This study uses a repeated-measures, longitudinal design to investigate associations between adversity exposure and learning-related cognitive control processes in the context of elevated depression (Aim 1). Adversity exposure and cognitive control will be examined as direct predictors of cognitive restructuring skill acquisition and skill retention over six-months; an indirect pathway from adversity to skill acquisition through cognitive control will also be examined (Aim 2). The study also includes exploration of key characteristics of adversity, namely the type (threat of harm versus deprivation of resources) and developmental timing of exposure, as distinct predictors of skill acquisition (exploratory Aim 3).

DETAILED DESCRIPTION:
ASSESSMENT: With verbal permission from the parent, both the interested parent and adolescent will complete an eligibility screener over the phone. The eligibility screener includes demographic information, psychiatric history, and current depression symptoms (self-report Patient Health Questionnaire-9, and the parent-report Children's Depression Inventory-2) to confirm that interested families meet initial inclusion criteria.

Baseline Assessment. A baseline assessment will be scheduled with all families. Informed consent and assent will be obtained prior to the start of any baseline assessment activities. A diagnostic interview (K-SADS-P/L) will be completed by a trained study staff member with each adolescent and their consenting parent. Diagnoses will be based on consensus ratings between adolescents and parents. Study staff will also administer the pediatric Columbia Suicide Severity Rating Scale, the Depression Rating Scale (embedded in K-SADS-P/L), and the Childhood Trauma Questionnaire.

The Wechsler Abbreviated Scale for Intelligence-II (WASI-II), the Cambridge Neuropsychological Test Automated Battery (CANTAB), and computerized tasks described in the outcome measures will be administered by a study staff member.

Self-report questionnaires will be administered to the parents and adolescents assessing peer victimization, community violence exposure, child and family demographics, stressful life events, food security, neglectful behaviors, social and cognitive stimulation during early childhood, discrimination, pubertal development, sleep behaviors, depression symptoms, and parent-child relationship quality.

Final study eligibility will be confirmed based on interviews and the WASI-II.

EXPERIMENTAL SKILL LEARNING AND ASSESSMENT Approximately one week following the baseline assessment (up to four weeks to allow for any scheduling difficulties) all participants will complete a 60-minute skill learning session. Prior to the experimental skills learning procedures, a study staff member will complete a brief (10-minute) interview with participants asking them to identify and describe a stressful event or interpersonal interaction from the past week. Participants will be asked to describe in detail how they coped with the event. Prompts will be given to elicit more detail when necessary. The purpose of the interview is to assess baseline cognitive restructuring skill use. After completing the interview, a trained study clinician will deliver the "Repairing Thoughts" skills module teaching cognitive restructuring from the "FIRST: Principal Based Approach to Evidence-based Psychotherapy" manual to the adolescent. The interview and the skills module may be audio and/or video recorded. Participants will be asked to practice their skill at home each day after the visit for the next week, and they will be sent an electronic daily survey to indicate whether they practiced.

Participants will be asked to complete a 90-minute, second session, one week later (up to three weeks to allow for any scheduling difficulties) to review the skill and practice in-vivo with the study clinician. After review and practice with the study clinician, a study staff member will meet with the adolescent participant to repeat the interview conducted during the first session.

As a part of this second skill learning session, a study staff member will introduce an in-vivo cognitive restructuring task to assess acquisition of the skill. Prior to the start of the in-vivo skill, resting-state continuous measurement of electrodermal activity (EDA; skin conductance), electrocardiogram (ECG), and respiration (RSP) will be collected at baseline. Study staff members (or the parent, if the adolescent prefers) will attach the electrodes and wireless transmitters (attached by velcro band to participants wrist and torso, on the exterior surface of clothing). After a baseline resting period, participants will be shown four brief film clips from movies or TV shows that have been extensively tested for reliably evoking negative emotions. Participants will be instructed to "watch" two clips, and to use cognitive restructuring to "reappraise" and reduce their emotional response during the remaining two clips (order counter-balanced). Continuous EDA, ECG, and RSP measurement will span the duration of the lab task and a three-minute recovery period that follows. The difference in physiological recovery between the "watch" and "reappraise" clips indexes cognitive restructuring ability.

Skill Retention Assessment. Participants will be sent online self-report surveys via the secure Qualtrics platform at 1-week, 3-months and 6-months follow-up. The interview conducted at pre- and post-skill learning sessions will also be repeated via phone at these timepoints. At 1-week follow-up, the online survey is a memory test for the cognitive restructuring skill. At 3-months follow-up and 6-months follow-up, self-report surveys will assess depression symptom levels, any psychotherapy or psychotropic medication services initiated since the last in-person visit, and the memory test for the cognitive restructuring skill. Adolescent participants will also re-complete the interview from the last in-person visit, conducted over the phone with study staff at all three follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages 12 years 0 months through 15 years 11 months at study enrollment
* Have clinically elevated depression symptom severity based a cut-off score of ≥ 7 on the Patient Health Questionnaire-9, verified by clinician ratings on the Depression Rating Scale.

Exclusion Criteria:

* Lifetime presence of a DSM-5 Psychotic or Autism Spectrum Disorder
* Lifetime presence of a neurological or serious medical condition
* Current DSM-5 diagnosis of substance abuse or dependence

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Cognitive Restructuring Skill Acquisition | Immediately post-intervention
  This primary outcome measure is an idiographic interview. A study staff member will conduct the brief idiographic interview asking participants to identify a stressful or negative event that occurred in the last week that elicited a negative emotional response. Participants will be asked to describe the event in detail, and then prompted to describe how they dealt with the event. Interviewer prompts to identify thoughts will be administered as needed. Interviews will be coded of cognitive restructuring strategies and a summary score of the amount and quality of cognitive restructuring components used will be calculated. Skill acquisition is defined as the summary score at post-intervention, controlling for summary scores at pre-intervention.
Cognitive Restructuring Skill Retention up to 6-months | Pre-intervention up to 6-months follow-up
  This primary outcome measure is an idiographic interview. A study staff member will conduct the brief idiographic interview asking participants to identify a stressful or negative event that occurred in the last week that elicited a negative emotional response. Participants will be asked to describe the event in detail, and then prompted to describe how they dealt with the event. Interviewer prompts to identify thoughts will be administered as needed. Interviews will be coded of cognitive restructuring strategies and a summary score of the amount and quality of cognitive restructuring components used will be calculated. Retention of the acquired skill is defined as the summary scores at each follow-up (1-week, 3-months, and 6 months post-intervention), controlling for summary scores at post-intervention.
Cognitive Restructuring Knowledge Test | Immediately post-intervention
  This outcome measure is a two-part self-report scale. The first component asks participants to describe all the steps to the cognitive restructuring skill and assesses knowledge of each component of the cognitive restructuring skill that participants learned. A total score is generated on a scale of 0-5 with higher scores indicating greater recall. The second component includes 10 multiple-choice items presenting hypothetical social scenarios with adolescents and participants are asked to rate the most likely interpretation of the situation. Correct answers reflect a use of cognitive restructuring to interpret ambiguous situations. A total score (0-10) is generated with higher scores indicating greater knowledge. This outcome measure is adapted from an existing self-report tool known as the Skill Acquisition Measure (SAM; Lindhiem and colleagues).
Biobehavioral sympathetic recovery | Immediately post-intervention
  This primary outcome is a measure of psychophysiological response in the form of electrodermal activity (EDA), also known as skin conductance, which captures autonomic arousal in the sympathetic nervous system. Biobehavioral recovery is defined as the slope of EDA recovery directly following the use of cognitive restructuring in response to a negative emotion induction (film clip).

SECONDARY OUTCOMES:
Biobehavioral parasympathetic regulation | Immediately post-intervention
  This secondary outcome measure captures autonomic recovery in the form of respiratory sinus arrhythmia (RSA), a measure of parasympathetic nervous system activity. RSA levels during a task where cognitive restructuring is used in response to negative emotion induction (film clip) is compared to RSA levels during a recovery period that immediately follows. RSA recovery is defined as the percent change in average RSA levels, comparing the emotion induction period to the recovery period.

OTHER OUTCOMES:
Self-reported depression symptom severity | Pre-intervention up to 6-months post-intervention
  The Mood and Feelings Questionnaire (MFQ) is a self-report questionnaire assessing youth depression symptoms in the last two weeks. Items are presented on a 3-point scale with ratings of 0=Not True, 1=Sometimes, and 2=True. A total sum score (range=0-66) is generated with higher scores indicating more severe symptoms. Reliability and validity of the scale has been well-established in existing psychometric research.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Vaughn-Coaxum, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data and protocol from this study will be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After study completion
Access Criteria: Open to public

REFERENCES:
- [Background] Weisz, J. R., & Bearman, S. K. (2020). Principle-Guided Psychotherapy for Children and Adolescents: The FIRST Program for Behavioral and Emotional Problems. Guilford Press.
- [Background] Gilman TL, Shaheen R, Nylocks KM, Halachoff D, Chapman J, Flynn JJ, Matt LM, Coifman KG. A film set for the elicitation of emotion in research: A comprehensive catalog derived from four decades of investigation. Behav Res Methods. 2017 Dec;49(6):2061-2082. doi: 10.3758/s13428-016-0842-x. PMID 28078572